CLINICAL TRIAL: NCT00147238
Title: A Validation Study of MR Lymphangiography Using SPIO, a New Lymphotropic Superparamagnetic Nanoparticle Contrast
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated at request of sponsor.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0003
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Results first posted 2010-01-27 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: Bladder Cancer; Genitourinary Cancer; Prostate Cancer
Keywords: Bladder Cancer; Genitourinary Cancer; Prostate Cancer; MR Lymphangiography; Ferumoxtran-10; SPIO; Ultra-small superparamagnetic agent iron oxide
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urogenital Neoplasms; Prostatic Neoplasms | interventions — ferumoxtran-10; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferumoxtran-10 MRI (Experimental): MR lymphangiography using Ferumoxtran-10 contrast agent.
  Interventions: Drug: Ferumoxtran-10 (USPIO); Procedure: MR lymphangiography
- MRI (Active Comparator): MR lymphangiography before injecting Ferumoxtran-10 contrast agent.
  Interventions: Procedure: MR lymphangiography

INTERVENTIONS:
Drug: Ferumoxtran-10 (USPIO) — Intravenous infusion of 2.6 mg/kg of ferumoxtran-10
  Other Names: MRI Contrast Agent; Ultra-small superparamagnetic oxide particles
  Arms: Ferumoxtran-10 MRI
Procedure: MR lymphangiography — First MRI examination before ferumoxtran-10 contrast injected and second MRI examination about 24 hours after injection of contrast agent, each MRI taking 20 minutes.
  Other Names: MRI; Magnetic Resonance Imaging

SUMMARY:
The goal of this clinical research study is to evaluate how well ferumoxtran-10, a new Magnetic Resonance Imaging (MRI) contrast agent, can detect cancer in the pelvic lymph nodes or malignant pelvic lymph nodes.

DETAILED DESCRIPTION:
The contrast agent, ferumoxtran-10, is made of ultra small iron oxide particles (USPIO). Once they are injected through vein, they are taken up mostly by liver, spleen, bone marrow, and lymph nodes. It takes about 24 - 36 hours to reach peak uptake in the lymph nodes. The ability of current imaging techniques to detect the lymph nodes disease is known to be less than perfect. Current techniques only use anatomic information (size). Previous studies have shown that this new contrast agent may be able to detect normal and abnormal lymph nodes, using MRI procedure, called MRI lymphangiogram. This new contrast agent is being evaluated to determine whether it can be used to detect normal and abnormal lymph nodes.

The study includes 2 parts. The first part will involve you receiving a MRI examination before the contrast is injected. The second part will involve you receiving a MRI examination about 24 hours after the injection. It will take about 20 minutes for each part.

If you are already scheduled to have a routine pelvic MRI, the first part of this study will be added at the end of the routine MRI. You will then be asked to return next day to complete the second part of the MRI. If you are not already scheduled to receive a MRI as part of your standard of care, you will come in to the MRI suite at M. D. Anderson and complete both parts over about a 24-hour interval.

You will be lying on the MRI examination table during the scanning. At the end of the first part of the study, the contrast will be infused slowly through vein over about 30 minutes in the recovery area. You will then be observed for 30 minutes to 2 hours, depending on your tolerance to the contrast agent. The images taken during the first part will be then be repeated 24-36 hours later. You will receive a follow-up telephone call from a member of the study staff on Day 3.

Once the second part of the MRI is performed, your participation in this study will be over.

This is an investigational study. This contrast agent is currently being evaluated by FDA and has not been approved yet. A total of 80 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed pelvic urological tumors, including prostate carcinomas, bladder carcinomas, and penile carcinomas.
2. Planned to have a surgical exploration or a laparoscopy for pelvic lymph node dissection/biopsy within 4 weeks.
3. Signed written consent and HIPAA authorization

Exclusion Criteria:

1. Contraindications for MRI
2. Claustrophobia, metals in the pelvis, previous pelvic surgery
3. Allergy or hypersensitivity to iron products, dextrans, iron-dextran complex
4. a. Prostate cancer: metastases demonstrated on preoperative imaging; prior hormonal therapy greater than 3 months; prior local therapy for prostate cancer b. Penile Cancer: prior systemic therapy for penile cancer; prior inguinal radiation c. Bladder Cancer: prior systemic therapy for bladder cancer (does NOT include intravesical chemotherapy or immunotherapy); prior pelvic radiation; history of partial cystectomy or prior pelvic lymph node dissection
5. Women of child-bearing potential. (Women who will be having hysterectomy as part of bladder surgery will not be excluded.)
6. Clinically documented or risk of primary or secondary iron overloading (e.g.History of thalassemia, sickle cell anemia, hereditary hemochromatosis, multiple transfusions with any reason)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-07; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haesun Choi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 08/24/05 through 06/12/06. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: A total of 10 patients enrolled prior to sponsor's request for early termination. Only 2 patients were evaluable for response therefore data will not be analyzed due to too small sample size.
Period: Overall Study
Arm/Group | Ferumoxtran-10 MRI Contrast Agent
Started | 10
Completed | 2
Not Completed | 8
Not completed — Inevaluable | 8

BASELINE CHARACTERISTICS:
Arm/Group | Ferumoxtran-10 MRI Contrast Agent
Number analyzed (Participants) | 10
Age Continuous [Mean (Full Range); unit: years] | 64 [55 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of MRI Per Patient
Description: Sensitivity of MRI on a per patient basis using two-sided McNemar test to detect differences in the sensitivities of two paired MR images (one with and one without ferumoxtran-10 contrast agent). Sensitivity of images written as percentage in decimal form: 0.0 (low) to 1.0 (high).
Time Frame: MRI without ferumoxtran-10 contrast and second repeated MRI with contrast agent within 24-36 hours of contrast injection, about 24 hours after first MRI
Population: Primary outcome measure was not assessed due to early study termination (e.g. patients did not receive assigned treatment).
Arm/Group | Ferumoxtran-10 MRI Contrast Agent
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 9 Months (September 2005-June 2006)
Arm/Group | Ferumoxtran-10 MRI Contrast Agent
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No